CLINICAL TRIAL: NCT00994227
Title: Clinicopathologic Findings for Macular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: hallym unuversity medical center, department of ophthalmology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-10-10
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Macular Disease
Keywords: electron microscopy; internal limiting membrane; macular disease; optical coherence tomography
MeSH Terms: conditions — Macular Degeneration | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery (Experimental)
  Interventions: Procedure: vitrectomy for macular disease

INTERVENTIONS:
Procedure: vitrectomy for macular disease — three-port pars plana vitrectomy was performed in each case using a vitreous cutter surrounded by a coaxial optic fiber connected to a xenon light source (Lausanne set, Oertli, Switzerland-developed at Jules Gonin, Lausanne, by Gonvers and Bovey). Separation of the posterior hyaloid membrane was performed when necessary. Visualization of the fundus was achieved with a special noncontact wide-angle viewing system 37 during vitrectomy and with a planoconcave contact lens for macular peeling. The MEM was peeled in the macular area using an end gripping forceps.
  Other Names: vitrectomy(DORC)

SUMMARY:
this study is to analyze and compare the ultrastructure of the retinal and vitreous plane of the epiretinal membrane and internal limiting membrane removed during macular surgery and to evaluate relation between the ultrastructure of the epiretinal membrane and internal limiting membrane and surgical outcomes.

DETAILED DESCRIPTION:
prospective, interventional study and includes patients who underwent vitrectomy,peeling of an epiretinal membrane and internal limiting membrane excision with or without intraoperative intraocular ICG injection.

Excised specimens were placed on a Millipore filter, fixed in a paraformaldehyde solution, and examined by light and transmission electron microscopy. Ultrathin sections were stained with uranyl acetate-lead citrate and inspected in a Zeiss EM electron microscope. The assessment was done in a blinded, masked fashion so that the clinicians who reviewed the histologic specimens

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent vitrectomy,peeling of an idiopathic MEM and ILM excision with or without intraoperative intraocular ICG injectio

Exclusion Criteria:

* the presence of macular hole or lamellar macular hole previous vitreoretinal surgery the presence of any other macular pathologic features potentially interfering with histologic results (such as diabetic retinopathy or age-related macular degeneration).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
spectral domain optical coherence tomography | baseline, 1week, 1month, 3 month
  The central 1mm subfield thickness the average macular thickness the inner nuclear layer thickness outer nuclear layer thickness outer plexiform layer thickness photoreceptor integrity ILM map RPE map
best corrected visual acuity | baseline, 1 month, 3 months
  logMAR

SECONDARY OUTCOMES:
electron microscopy finding of internal limiting membrane | during operation
visual field | baseline, postoperative 1 months, 3 months
  humpley visual field
preferential hyperacuity perimeter | baseline, postoperative 1 months, 3 months
  ForeseePHP 2.05; Notal Vision, Tel Aviv, Israel

CONTACTS AND LOCATIONS:
Locations (1):
- JiWon Lim, Seoul, South Korea

REFERENCES:
- [Derived] Lim JW, Kim HK, Cho DY. Macular function and ultrastructure of the internal limiting membrane removed during surgery for idiopathic epiretinal membrane. Clin Exp Ophthalmol. 2011 Jan;39(1):9-14. doi: 10.1111/j.1442-9071.2010.02377.x. PMID 20662848